CLINICAL TRIAL: NCT03736252
Title: Effectiveness of a Neoprene CMC Joint Orthosis for Pain, Function, and Patient Satisfaction
Brief Title: Effectiveness of a Neoprene CMC Joint Orthosis
Acronym: Carpometacar
Status: Completed | Type: Observational
Sponsor: Gannon University (Other)
Responsible Party: Principal Investigator, Kristin Valdes, Assistant Professor, Gannon University
Other Study IDs: GUIRB-2018-8-66
Record Dates: First submitted 2018-11-07; First posted 2018-11-09 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: CMC
Keywords: Orthosis; Pain; Function
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Orthosis provision — Hely and Weber CMC controller

SUMMARY:
Patients will be gathered via convenience sample from a hand therapy clinic. They will be provided with a neoprene commercially available orthosis free of charge. Baseline pain and function will be assessed using the VAS and Functional Index of Hand Arthropathies. Four weeks later, pain, function, and patient satisfaction with the device will be gathered using the Quebec User Evaluation of Assistive Technology questionnaire.

DETAILED DESCRIPTION:
Patients with the diagnosis of carpometacarpal osteoarthritis that are receiving hand therapy will be recruited for the study. Baseline measurements will include usual pain over the past week, current pain, and worst pain experienced over the past week using the VAS pain scale. Hand function will be assessed using the Functional Index of Hand Arthropathies measure. The patients will be provided with a free neoprene hand orthosis (Hely and Weber CMC controller). They will be instructed to wear the device as needed for pain. After 1 month, the investigators will call the patient to assess pain, function, and satisfaction with the device using the Quebec User Evaluation of Assistive Technology Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* CMC OA of either thumb with pain

Exclusion Criteria:

* CMC arthroplasty
* recent surgery
* dementia
* no pain at CMC joint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with painful CMC OA
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Pain using the Visual Analog Scale (VAS) scale | 1 month
  Pain measured with VAS pain scale, measured from 1-10. 1 is the best and 10 is the worst

SECONDARY OUTCOMES:
Hand osteoarthritis Function | 1 month
  Function measured with FIHOA.The FIHOA assesses hand OA-related functional impairment scoring from 0 (no functional impairment) to 30 points (maximal impairment).The total score ranges from 0 to 30, with a validated threshold of 5 able to distinguish between symptomatic and not symptomatic patients or controls.
Patient satisfaction with device: Quebec User Evaluation of Satisfaction with Assistive Technology | 1 month
  Measured with QUEST scale. The Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) is a 12-item outcome measure that assesses user satisfaction with two components, Device and Services. Scores of 1 indicate dissatisfaction and scores of 5 indicate high satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Gannon University, Ruskin, Florida, United States

IPD SHARING:
Plan to Share IPD: No